CLINICAL TRIAL: NCT01290757
Title: Bioequivalence of Two Different Capsule Types of 150 mg Dabigatran Etexilate Made From Two Different Drug Product Batches, Following Oral Administration in Healthy Male and Female Volunteers (Open-label, Randomised, Single Dose, Replicate Design in a Two Treatments, Four Periods Crossover Phase I Study)
Brief Title: Bioequivalence of Two Different Capsule Types of Dabigatran
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.117; 2010-022966-28 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-02-02; First posted 2011-02-07 (Estimated); Results first posted 2012-06-29 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (2):
- Dabigatran etexilate 150 mg (T) (Experimental): Capsugel (T), oral administration
  Interventions: Drug: Dabigatran etexilate
- Dabigatran etexilate 150 mg (R) (Experimental): Qualicaps (R), oral administration
  Interventions: Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: Dabigatran etexilate — 150 mg Capsugel (T)
  Arms: Dabigatran etexilate 150 mg (T)
Drug: Dabigatran etexilate — 150 mg Qualicaps (R)
  Arms: Dabigatran etexilate 150 mg (R)

SUMMARY:
The objective of this Phase I trial is to demonstrate the bioequivalence of two capsules of dabigatran etexilate made from two different drug product batches.

The reference batch is dabigatran etexilate hard capsules 150 mg using the currently approved capsule shell (Qualicaps). The test batch is dabigatran etexilate 150 mg hard capsules using a new capsule shell (Capsugel). The test batch is the drug product intended for future commercial use.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
2. Age =21 and = 55 years
3. Body Mass Index (BMI) =18.5 and BMI = 29.9 kg/m^2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion criteria:

1. Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Clinically relevant surgery of gastrointestinal tract or evidence of significant gastrointestinal motility problems that could affect absorption of the drug
3. Diseases of the central nervous system (included but not limited to any kind of seizures, stroke or psychiatric disorders) within the past 6 month
4. Any history or evidence of blood dyscrasia, hemorrhagic diathesis, severe thrombocytopenia, cerebrovascular hemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with hemorrhagic tendencies
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy in particular to study drug or its excipients) which is deemed relevant to the trial as judged by the investigator
8. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
9. Alcohol abuse (more than 20 g/day)
10. Drug abuse
11. Any laboratory value outside the reference range that is of clinical relevance (especially hemoglobin, thrombocytes, prothrombin time (PT) and Activated Partial Thromboplastin Time (Measure of the clotting time) (aPTT) or positive drug or virus screening
12. Planned surgeries within four weeks following the end-of study examination
13. Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding within 14 days before or after end-of study examination

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.117.1 Boehringer Ingelheim Investigational Site, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this crossover study, subjects were randomly assigned to one of the 2 sequences, with 2 treatment arms. In general terms, Ref-Test-Ref-Test and Test-Ref-Test-Ref. The aim was bioequivalence comparing (Ref) Dabigatran 150mg in the currently approved capsule shell (Qualicaps) to the test of Dabigatran 150mg in a new shell (Capsugel).
Groups:
- Sequence: Qualicaps - Capsugel - Qualicaps - Capsugel: Dabigatran 150mg in currently approved Qualicaps, followed by Dabigatran 150mg in new Capsugel, followed by Dabigatran 150mg in currently approved Qualicaps, followed by Dabigatran 150mg in new Capsugel (RTRT)
- Sequence: Capsugel - Qualicaps - Capsugel - Qualicaps: Dabigatran 150mg in new Capsugel, followed by Dabigatran 150mg in currently approved Qualicaps, followed by Dabigatran 150mg in new Capsugel, followed by Dabigatran 150mg in currently approved Qualicaps (TRTR)
Period: Overall Study
Arm/Group | Sequence: Qualicaps - Capsugel - Qualicaps - Capsugel | Sequence: Capsugel - Qualicaps - Capsugel - Qualicaps
Started | 90 | 90
Completed | 88 | 88
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set includes all patients who received at least one study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence: Qualicaps - Capsugel - Qualicaps - Capsugel | Sequence: Capsugel - Qualicaps - Capsugel - Qualicaps | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (10.1) | 39.4 (9.1) | 39.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0 to tz (AUC0-tz) of Total Dabigatran
Description: Area under the concentration-time curve of total dabigatran in plasma from time 0 to the time of the last quantifiable data point, adjusted for treatment, period and sequence (all fixed effects), and random subject effect.
Time Frame: 60 hours
Population: This subject set, the pharmacokinetic set (PKS), includes all subjects of the treated set who provide at least one evaluable observation for at least one of the three PK endpoints of total dabigatran, which is obtained in a period without important protocol violations relevant to the evaluation of bioequivalence.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Capsugel: Dabigatran 150mg in new Capsugel
- Qualicaps: Dabigatran 150mg in currently approved Qualicaps
Arm/Group | Capsugel | Qualicaps
Number analyzed (Participants) | 179 | 180
ng*hr/mL | 1147.64 (32.32) | 908.48 (49.83)
Statistical Analysis 1: Comparison: Capsugel vs Qualicaps; Capsugel minus Qualicaps; Test type: Non-Inferiority or Equivalence — Bioequivalence (BE). Scaled average BE is rejected, if the calculated upper 95% confidence limit of the linearized criterion is positive; Mixed Models Analysis; Upper 95% CI of the linearized criterion = -0.082 — Linearized regulatory criterion according to Tothfalusi et al (Pharmaceutical Research, 2001). The square of the difference in treatment responses divided by within-subject variance of the reference formulation minus square of ln(1.25)/0.25
Statistical Analysis 2: Comparison: Capsugel vs Qualicaps; Capsugel vs Qualicaps; Test type: Non-Inferiority or Equivalence — Bioequivalence (BE). Bioequivalence is accepted if 90% confidence interval lies within the common BE margins (80% and 125%); Mixed Models Analysis; Adjusted geometric mean ratio (%) = 126.33, 90% CI [119.45 to 133.60]

2. Primary Outcome: Maximum Measured Concentration (Cmax) of Total Dabigatran in Plasma
Description: Adjusted for treatment, period and sequence (all fixed effects), and random subject effect.
Time Frame: 60 hours
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Capsugel | Qualicaps
Number analyzed (Participants) | 179 | 180
ng/mL | 134.44 (31.10) | 107.13 (49.67)
Statistical Analysis 1: Comparison: Capsugel vs Qualicaps; Capsugel minus Qualicaps; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Upper 95% CI of the linearized criterion = -0.085 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Capsugel vs Qualicaps; Capsugel vs Qualicaps; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; Adjusted geometric mean ratio (%) = 125.49, 90% CI [118.69 to 132.67]

3. Secondary Outcome: Area Under the Curve 0 to Infinity (AUC0-∞) of Total Dabigatran.
Description: Area under the concentration-time curve of total dabigatran in plasma over the time interval from 0 extrapolated to infinity. Adjusted for treatment, period and sequence (all fixed effects), and random subject effect.
Time Frame: 60 hours
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Capsugel | Qualicaps
Number analyzed (Participants) | 179 | 180
ng*hr/mL | 1175.05 (30.81) | 941.99 (46.53)
Statistical Analysis 1: Comparison: Capsugel vs Qualicaps; Capsugel vs Qualicaps; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; Adjusted geometric mean ratio (%) = 124.74, 90% CI [118.32 to 131.51]

4. Secondary Outcome: AUC0-tz of Free Dabigatran.
Description: Area under the concentration-time curve of free dabigatran in plasma from time 0 to the time of the last quantifiable data point. Adjusted for treatment, period and sequence (all fixed effects), and random subject effect.
Time Frame: 60 hours
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Capsugel | Qualicaps
Number analyzed (Participants) | 179 | 180
ng*hr/mL | 856.31 (33.15) | 678.43 (50.85)
Statistical Analysis 1: Comparison: Capsugel vs Qualicaps; Capsugel vs Qualicaps; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; Adjusted geometric mean ratio (%) = 126.22, 90% CI [119.36 to 133.47]

5. Secondary Outcome: Cmax of Free Dabigatran in Plasma.
Description: Adjusted for treatment, period and sequence (all fixed effects), and random subject effect.
Time Frame: 60 hours
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Capsugel | Qualicaps
Number analyzed (Participants) | 179 | 180
ng/mL | 106.66 (31.34) | 85.12 (50.33)
Statistical Analysis 1: Comparison: Capsugel vs Qualicaps; Capsugel vs Qualicaps; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; Adjusted geometric mean ratio (%) = 125.30, 90% CI [118.42 to 132.59]

6. Secondary Outcome: AUC0-∞ of Free Dabigatran.
Description: Area under the concentration-time curve of free dabigatran in plasma over the time interval from 0 extrapolated to infinity. Adjusted for treatment, period and sequence (all fixed effects), and random subject effect.
Time Frame: 60 hours
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Capsugel | Qualicaps
Number analyzed (Participants) | 179 | 180
ng*hr/mL | 888.86 (31.20) | 714.01 (47.16)
Statistical Analysis 1: Comparison: Capsugel vs Qualicaps; Capsugel vs Qualicaps; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; Adjusted geometric mean ratio (%) = 124.49, 90% CI [118.11 to 131.21]

ADVERSE EVENTS:
Time Frame: Approximately 7 days
Groups:
- Qualicaps: Dabigatran 150mg in Qualicaps
- Capsugel: Dabigatran 150mg in Capsugel
Arm/Group | Qualicaps | Capsugel
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180
Other Adverse Events (participants affected / at risk) | 37/180 | 34/180
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Qualicaps (N=180) | Capsugel (N=180)
Headache (Nervous system disorders) | 37 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.